CLINICAL TRIAL: NCT06830135
Title: A Multifaceted Telehealth Approach to Enhancing Glycemic Control and Reducing Readmissions in a Diverse Diabetic Population: A Randomized Control Trial
Brief Title: Telehealth Approach to Enhancing Glycemic Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: White Plains Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WPH IRB: 2025-16585
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; continuous glucose monitoring; remote patient monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm -standard of care (No Intervention)
- Intervention Arm (Experimental): Continuous glucose monitoring, remote patient monitoring for 90 days
  Interventions: Device: Continues glucose monitoring with remote glucose monitoring for 90 days

INTERVENTIONS:
Device: Continues glucose monitoring with remote glucose monitoring for 90 days — CGM + RPM
  Arms: Intervention Arm

SUMMARY:
This study evaluates whether the use of a Continuous Glucose Monitoring (CGM) device combined with a Remote Patient Monitoring (RPM) program can improve blood sugar control and reduce hospital visits among patients with poorly controlled diabetes who have recently been discharged from the hospital.

The study, led by White Plains Hospital (WPH) Cares, will follow 208 patients for 90 days after their discharge. Half of the participants will receive standard care, while the other half will receive a Dexcom G7 CGM device along with support from trained nurses who will monitor their glucose readings daily. The goal is to determine whether this approach helps lower Hemoglobin A1c (HbA1c) levels, reduces hospital readmissions, and improves overall health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Discharged Home from the WPH Inpatient Setting A1c >= 8.0 within 90 days of discharge >= 18 Years of Age Lives within Westchester County

Exclusion Criteria:

* <18 Years of Age Patient With Documented Cognitive Impairment or Decisional Incapacity Pregnant or Plans to Become Pregnant in 6 Months Discharge Disposition of Short-term or Long-term Care Facility, Assisted Living Facility, Group Home, Against Medical Advice/Eloped, or Home Hospice Patient or Caregiver Unable to Check Glucose at Home Using a Home Glucometer Lives Outside Westchester County

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 90 days

SECONDARY OUTCOMES:
30 days hospital readmissions | 30 days
Overall healthcare utilization | 90 days
Acute care visits related to abnormal glucose reading | 30 days

OTHER OUTCOMES:
Percentage of Patients Enrolled in the Program | 2 years
Changes in Medical Glucose Readings | 7 day
Equity in Program Participation | 2 years
  (% of Participants Who Are Hispanic, African American, or Uninsured)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen JA, Scoggins D, Michaud T, Wan N, Wen M, Su D. Racial Disparities in Diabetes Management Outcomes: Evidence from a Remote Patient Monitoring Program for Type 2 Diabetic Patients. Telemed J E Health. 2021 Jan;27(1):55-61. doi: 10.1089/tmj.2019.0280. Epub 2020 Apr 17. PMID 32302521
- [Background] Elsener M, Santana Felipes RC, Sege J, Harmon P, Jafri FN. Telehealth-based transitional care management programme to improve access to care. BMJ Open Qual. 2023 Nov;12(4):e002495. doi: 10.1136/bmjoq-2023-002495. PMID 37940335
- [Background] Greenwood DA, Young HM, Quinn CC. Telehealth Remote Monitoring Systematic Review: Structured Self-monitoring of Blood Glucose and Impact on A1C. J Diabetes Sci Technol. 2014 Mar;8(2):378-389. doi: 10.1177/1932296813519311. Epub 2014 Feb 21. PMID 24876591
- [Background] Salehi S, Olyaeemanesh A, Mobinizadeh M, Nasli-Esfahani E, Riazi H. Assessment of remote patient monitoring (RPM) systems for patients with type 2 diabetes: a systematic review and meta-analysis. J Diabetes Metab Disord. 2020 Jan 10;19(1):115-127. doi: 10.1007/s40200-019-00482-3. eCollection 2020 Jun. PMID 32550161
- [Background] Pal K, Eastwood SV, Michie S, Farmer A, Barnard ML, Peacock R, Wood B, Edwards P, Murray E. Computer-based interventions to improve self-management in adults with type 2 diabetes: a systematic review and meta-analysis. Diabetes Care. 2014 Jun;37(6):1759-66. doi: 10.2337/dc13-1386. PMID 24855158
- [Background] Boye KS, Thieu VT, Lage MJ, Miller H, Paczkowski R. The Association Between Sustained HbA1c Control and Long-Term Complications Among Individuals with Type 2 Diabetes: A Retrospective Study. Adv Ther. 2022 May;39(5):2208-2221. doi: 10.1007/s12325-022-02106-4. Epub 2022 Mar 22. PMID 35316502
- [Background] Steinhubl SR, Muse ED, Topol EJ. The emerging field of mobile health. Sci Transl Med. 2015 Apr 15;7(283):283rv3. doi: 10.1126/scitranslmed.aaa3487. PMID 25877894
- [Background] Rodriguez-Gutierrez R, Herrin J, Lipska KJ, Montori VM, Shah ND, McCoy RG. Racial and Ethnic Differences in 30-Day Hospital Readmissions Among US Adults With Diabetes. JAMA Netw Open. 2019 Oct 2;2(10):e1913249. doi: 10.1001/jamanetworkopen.2019.13249. PMID 31603490
- [Background] Soh JGS, Wong WP, Mukhopadhyay A, Quek SC, Tai BC. Predictors of 30-day unplanned hospital readmission among adult patients with diabetes mellitus: a systematic review with meta-analysis. BMJ Open Diabetes Res Care. 2020 Aug;8(1):e001227. doi: 10.1136/bmjdrc-2020-001227. PMID 32784248
- [Background] Centers for Disease Control and Prevention. National Diabetes Statistics Report, 2020. Atlanta, GA, Centers for Disease Control and Prevention, U.S. Department of Health and Human Services, 2020, p. 12-15
- [Background] U.S. Census Bureau. (2022). How has Westchester County's Racial and Ethnic Populations Changed. USA Facts. https://usafacts.org/data/topics/people-society/population-and-demographics/our-changing-population/state/new-york/county/westchester-county/. Accessed 12/9/2023.
- [Background] Westchester Community Foundation (2018) Health: Diabetes Mortality, by Race/Ethnicity. Westchester Index; An Initiative of Westchester County Foundation. https://westchesterindex.org/health/diabetes-mortality-by-race-ethnicity
- [Background] Smithwick, K. (n.d.). Diabetes Mortality, by race/ethnicity. Westchester Index. Retrieved November 3, 2022, from https://westchesterindex.org/health/diabetes-mortality-by-race-ethnicity.
- [Background] NY DOH, (2018). Percentage of Adults with Diagnosed Diabetes, by county, New York State, BRFSS 2018. New York Health. https://www.health.ny.gov/statistics/prevention/injury_prevention/information_for_action/docs/2021-01_ifa_report.pdf
- [Background] CDC. (n.d.). Diabetes State Burden Toolkit. Center for Disease Control and Prevention. https://nccd.cdc.gov/Toolkit/DiabetesBurden/TotalCost. Accessed 12/8/2023.
- [Background] American Diabetes Association. (2021). The Burden of Diabetes in New York. American Diabetes Association. https://www2.diabetes.org/sites/default/files/2021-11/ADV_2021_State_Fact_sheets_New%20York_rev.pdf
- [Background] CDC. (n.d.). Diabetes Data and Statistics. Center for Disease Control and M/edicine. Diabetes Data and Statistics. CDC. https://www.cdc.gov/diabetes/data/statistics-report/index.html. Accessed 12/7/2023